CLINICAL TRIAL: NCT06461624
Title: Clinical Trial of Autologous GPC3 CAR-T Cells (CBG166) Therapy for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Carbiogene Therapeutics Co. Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRKBY-201
Record Dates: First submitted 2024-06-05; First posted 2024-06-17 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: GPC3; Chimeric antigen receptor T cell; Adoptive cell therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPC3 CAR-T (CBG166) (Experimental)
  Interventions: Biological: anti-GPC3 CAR-T

INTERVENTIONS:
Biological: anti-GPC3 CAR-T — All subjects were intravenous administrated with CBG166.
  Other Names: CBG166 CAR-T

SUMMARY:
A phase I clinical study of 4th generation chimeric antigen receptor T Cells targeting glypican-3 ( CAR-GPC3 T Cells) in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a single-arm, dose-escalation, open, exploratory clinical study to evaluate the safety and tolerability, preliminary efficacy and PK/PD characteristics of GPC3 CAR-T cells in the treatment of advanced hepatocellular carcinoma.

Primary objectives: To evaluated the safety of GPC3 CAR-T cells in patients with advanced hepatocellular carcinoma.

Secondary objectives:To evaluate the preliminary efficacy and PK/PD characteristics of CBG166.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years, male or female;
* Subjects voluntarily participated in the research and signed the Informed Consent Form (ICF) by themselves or their guardians;
* Unresectable stage B or C HCC according to the Barcelona Clinic Liver Cancer (BCLC) staging. In case of stage B, the subject must have disease progression following surgery or local treatment, or be unsuitable for surgery or local treatment;
* Subjects have previously received at least one systemic treatment regimen (including but not limited to targeted therapy, immunotherapy or chemotherapy) with disease progression determined by imaging during or after treatment;
* Cirrhosis status Child-Pugh score:≤7;
* Intrahepatic lesions were confirmed by imaging examination (arterial phase enhancement) within 28 days before the start of treatment. According to the RECIST1.1, there was at least one target lesion that could be stably evaluated;
* Expected survival time > 12 weeks;
* Expression of GPC3 demonstrated by immunohistochemistry (IHC)
* ECOG Performance Status score: 0 to 1 point;
* Subjects should have adequate organ function;
* Subjects should be HBsAg negative. Subjects with positive HBsAg or positive HBcAb are required to have HBV-DNA <2000 IU/ml;
* The blood pregnancy test of female subjects of childbearing age should be negative within 7 days before cell therapy and not during lactation; Female or male subjects of childbearing age need to take efficient tools or drug contraceptive measures during the whole research process or within one year after CAR-T cell transfusion (What happens later shall prevail);

Exclusion Criteria:

* Subjects with completely resectable liver tumors or who are eligible for liver transplantation;
* Pregnant or lactating women;
* Active bacterial or fungal infections within 72 hours prior to gonorrhea clearance (excluding subjects who have no evidence of active infections and antibiotics are not on the prohibited drug list, and continue to use prophylactic antibiotics, antifungal drugs, or antiviral drugs);
* Patients who had received systemic steroids equivalent to > 15 mg/day prednisone within 2 weeks before apheresis, except those who had recently used or are currently using inhaled steroids;
* Before apheresis, Hb < 80 g/L, ANC < 1.0 × 109 /L or PLT < 60 × 109 /L;
* Current clinically significant ascites, which is defined as ascites that are physically positive or require intervention (e.g., puncture or medication) for control (those whose imaging result shows ascites requiring no intervention may be included);
* Imaging results:≥50% of the liver is replaced by tumor or portal vein main tumor thrombus, or tumor thrombus invasion of mesenteric vein / inferior vena cava;
* Previous or present hepatic encephalopathy;
* Active brain metastasis;
* Subjects with a history of organ transplantation or waiting for organ transplantation (including liver transplantation);
* Any of the following situations exist: Hepatitis B core antibody (HBcAb) positive and hepatitis B virus (HBV) DNA in peripheral blood isperipheral blood hepatitis B virus (HBV) DNA ≥ 2000 IU/mL. Hepatitis C virus (HCV) antibody positive and HCV RNA positive. Human immunodeficiency virus (HIV) antibody positive. Syphilis test positive.
* Other serious medical conditions that may limit the patient's participation in this trial;
* Subjects who received anti-tumor therapy within 2 weeks prior to apheresis, or who received any investigational drug or systemic anti-tumor therapy within 28 days (or 5 half-lives of the drug, whichever is more appropriate in the judgment of the investigator) prior to signing the informed consent form;
* Prior treatment with any therapy that is targeted to GPC3;
* At the time of signing the informed consent, toxicity caused by previous PD-1/PD-L1 treatment had not returned to grade 1 or baseline levels, except for hair loss and pigmentation;
* Other uncured malignant tumors in the past 5 years or at the same time, except for cervical cancer in situ and basal cell carcinoma of the skin;
* According to the investigators' evaluation, patients are unable or unwilling to comply with the requirements of the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Within 28 days of CAG166 infusion
  Describe the adverse events of limiting further increases in the dose of CBG166.
Adverse events | Within 24 months after the treatment
  Describe adverse events (AEs) and serious adverse events (SAEs) that are "likely" or "definitely" related to the study treatment that occur at any time of 24 months after treatment.
Maximum tolerated dose | From enrollment of the first subject to completion of follow-up of the last subject (up to 3 years)
  Determine the optimal agent for CBG166 CAR-T at maximum tolerated dose.

SECONDARY OUTCOMES:
Effectiveness evaluation | At weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  Objective response rate by RECIST 1.1
Effectiveness evaluation | The efficacy is evaluated at weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  Progression-free survival by RECIST 1.1
Effectiveness evaluation | The efficacy is evaluated at weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  Duration of response by RECIST 1.1
Effectiveness evaluation | The efficacy is evaluated at weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  Time to response by RECIST 1.1
Effectiveness evaluation | The efficacy is evaluated at weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  Disease control time by RECIST 1.1
Pharmacokinetic evaluation | Within 24 months after the treatment
  Detect duration and expansion of CAR-T cells in vivo
Pharmacodynamic evaluation | At weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  The copy number of HBV DNA in blood
Pharmacodynamic evaluation | At day 1, 4, 7, 15 and 21 and weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  The serum level of IFN-α2
Pharmacodynamic evaluation | At weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  The serum level of TGF-β
Pharmacodynamic evaluation | At weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  The serum level of soluble AFP
Pharmacodynamic evaluation | At weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  The serum level of soluble GPC3
Pharmacodynamic evaluation | At day 1, 4, 7, 15 and 21 and weeks 4, 8, and 18 and months 3, 4, 6, 9, 12, 15, 18 and 24 after cell infusion
  The serum levels of cytokine/chemokin

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang
  - the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No